CLINICAL TRIAL: NCT03383874
Title: A Probiotic Intervention to Prevent Relapse Following Hospitalization for Mania
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Sherwood Brown, MD, PhD, Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU 082017-045
Record Dates: First submitted 2017-12-19; First posted 2017-12-26 (Actual); Results first posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Mania (Neurotic)
Keywords: Probiotic, bipolar disorder, schizoaffective disorder, mania
MeSH Terms: conditions — Mania; Bipolar Disorder; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants will receive capsules containing placebo for 24-weeks.
  Interventions: Other: Placebo
- Probiotic-Probio-Tec BG-VCap-6.5 (Experimental): Participants will receive capsules containing approximately 10^9 colony forming units of the probiotic organisms, Lactobacillus GG and Bifidobacteria lactis strain Bb12 for 24-weeks.
  Interventions: Combination Product: Probio-Tec BG-VCap-6.5

INTERVENTIONS:
Combination Product: Probio-Tec BG-VCap-6.5 — The product under investigation is a probiotic containing two microorganisms (Lactobacillus rhamnosus, LGG® and Bifidobacterium animalis subsp. lactis, BB-12®, referred to as LGG® and BB-12®, respectively) and is offered commercially as "Probio-Tec BG-VCap-6.5". This composition is formulated to contain a minimum of 1 billion (1.0 x 10^9) CFU (Colony Forming Units) per dose (capsule), including equal numbers of the two strains; i.e. 0.5 x 10^9 CFU of each of LGG® and BB-12® at the time of manufacture. The product will be administered orally.
  Arms: Probiotic-Probio-Tec BG-VCap-6.5
Other: Placebo — This placebo is made almost identically to the Probio-Tec but without active microorganisms.
  Arms: Placebo

SUMMARY:
This will be a 24-week, randomized, double-blind, placebo-controlled trial of adjunctive probiotic therapy in 66 persons hospitalized with a manic or mixed episode. The active study compound will consist of capsules containing approximately 10^9 colony forming units of the probiotic organisms, Lactobacillus GG and Bifidobacteria lactis strain Bb12. The dose has been selected because it has been used safely in other probiotic trials, was well-tolerated by the participants in two previous trials of individuals with schizophrenia or mania, and was utilized in the original trial on which this replication is based. This dose is higher than that available in most commercially-sold health food supplements. Following hospital discharge, participants will be randomized to receive adjunctive probiotic or placebo for a 24 week period. It is anticipated that of the 66 participants randomized, ~50 (75%) will complete the full 24 weeks of the study. The primary outcome is relapse, defined as re-hospitalization (e.g., admission to an inpatient unit) for psychiatric symptoms following a previous hospital discharge by at least 2 weeks. The occurrence of new mood episodes, the severity of psychiatric symptoms, and any changes in cognitive test scores over the course of the study will also be evaluated. Changes in the levels of inflammatory markers as well as changes in gut microbiota will be evaluated at three time intervals over the course of the study.

DETAILED DESCRIPTION:
Primary Aim 1. To determine if adjunctive probiotic administration can reduce relapse for participants first hospitalized for mania. Hypothesis: Participants receiving adjunctive probiotic microorganisms vs. adjunctive placebo will have a lower rate of relapse as defined by a re-hospitalization (e.g., admission to an inpatient unit) during the 24 week study period.

Secondary Outcomes. The number of new mood episodes, the severity of psychiatric symptoms, and changes in cognitive scores over the 24 week study period will be evaluated.

Exploratory Aim 1. To study the effect of probiotic therapy in lowering the levels of inflammatory markers following an acute episode of mania. Hypothesis: Participants receiving adjunctive probiotic microorganisms vs. adjunctive placebo will have reduced levels of antibodies to casein, gliadin, and the NMDA receptor, and reduced levels of C-Reactive protein and the cytokine TNF alpha following 24 weeks of probiotic therapy.

Exploratory Aim 2. To evaluate changes in the gut microbiota following probiotic administration. Hypothesis: Probiotic administration will enrich the gut microbiota of participants with the given microorganisms and these changes may correlate to changes in the peripheral inflammatory markers being measured.

ELIGIBILITY:
Inclusion Criteria:

* Capacity for written informed consent
* Currently (or within the last 3 weeks) admitted to inpatient hospital for symptoms of mania.
* Primary Axis I diagnosis (DSM-5) at time of admission of bipolar I (single manic episode, most recent episode manic, or most recent episode mixed) OR schizoaffective disorder, bipolar type (manic or mixed state).
* Proficient in the English language.
* Available to attend follow-up visits.

Exclusion Criteria:

* Substance- or medically-induced symptoms of mania at time of assessment.
* HIV infection or other immunodeficiency condition (such as receiving cancer chemotherapy).
* A serious medical condition that affects brain or cognitive functioning (e.g., epilepsy, serious head injury, concussion involving loss of consciousness, brain tumor, or other neurological disorder). Note that Hepatitis-C is not an exclusion criterion unless the participant has an acute infection.
* Poorly controlled comorbid medical condition.
* Major surgery in the last year.
* History of weight loss surgery.
* Diagnosis of Intellectual Disability or history of severe learning disorder.
* Diagnosis of alcohol or substance use disorder (moderate/severe) according to DSM-5 criteria within the last 3 months, or has a positive drug toxicity screen proximate to the time of recruitment.
* History of IV drug use.
* Participated in any investigational drug trial in the past 30 days.
* Abnormal electrolyte levels.
* AST and ALT > 3 times upper limit of normal.
* Pregnant, breastfeeding, or planning to become pregnant during the study period.
* Documented celiac disease (as such persons should be on a gluten-free diet as this is the standard care). Of note, we are not limiting the study to individuals with elevated levels of gliadin or casein antibodies as we intend to look at these levels as a predictor of response.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2018-09-06 (Actual); Primary Completion 2024-09-23 (Actual); Study Completion 2024-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherwood Brown, MD, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Psychoneuroendocrine Research Program, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Probiotic-Probio-Tec BG-VCap-6.5
Started | 36 | 31
Completed | 20 | 25
Not Completed | 16 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Probiotic-Probio-Tec BG-VCap-6.5 | Total
Number analyzed (Participants) | 36 | 31 | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 2
  Between 18 and 65 years | 35 | 30 | 65
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.97 (17.08) | 32.29 (10.18) | 33.19 (12.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 18 | 35
  Male | 19 | 13 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 8 | 12 | 20
  White | 25 | 17 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 5 | 19
  Not Hispanic or Latino | 22 | 26 | 48
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Rate of Relapse
Description: 'Relapse' is defined as re-hospitalization (e.g., admission to an inpatient unit) for psychiatric symptoms following a previous hospital discharge by at least 2 weeks. The rate of relapse was calculated by dividing the number of re-hospitalizations per group (i.e., Placebo, Probiotic) by the number of participants per group so the unit is re-hospitalizations/participant.
Time Frame: 24 weeks
Measure: Number; unit: Proportion of Participants
Arm/Group | Placebo | Probiotic-Probio-Tec BG-VCap-6.5
Number analyzed (Participants) | 36 | 31
Proportion of Participants | .11 | .13

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Placebo | Probiotic-Probio-Tec BG-VCap-6.5
All-Cause Mortality (participants affected / at risk) | 1/36 | 0/31
Serious Adverse Events (participants affected / at risk) | 3/36 | 1/31
Other Adverse Events (participants affected / at risk) | 20/36 | 20/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=36) | Probiotic-Probio-Tec BG-VCap-6.5 (N=31)
Hospitalization due to Manic Symptoms (Psychiatric disorders) | 1 (2) | 1 (1)
Death due to Surgical Complication (Surgical and medical procedures) | 1 (1) | 0 (0)
Suicide Attempt (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=36) | Probiotic-Probio-Tec BG-VCap-6.5 (N=31)
Bloating (Gastrointestinal disorders) | 5 (5) | 1 (1)
Common Cold (Infections and infestations) | 3 (3) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 10 (14) | 7 (7)
Flatulence (Gastrointestinal disorders) | 3 (4) | 1 (1)
Stomach Discomfort (Gastrointestinal disorders) | 2 (3) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Increased Appetite (Gastrointestinal disorders) | 1 (1) | 3 (3)
Increased Frequency of Bowel Movements (Gastrointestinal disorders) | 0 (0) | 3 (5)
Indigestion (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Weight Gain (Metabolism and nutrition disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-18): https://cdn.clinicaltrials.gov/large-docs/74/NCT03383874/Prot_SAP_000.pdf
  • Informed Consent Form (2024-03-18): https://cdn.clinicaltrials.gov/large-docs/74/NCT03383874/ICF_001.pdf